CLINICAL TRIAL: NCT03497338
Title: the Efficacy and Safety of New Anticoagulation Strategies of Maintain Normal Clot Rate to Prevent Hemorrhage While VV-ECMO
Brief Title: New Anticoagulation Strategies of VV-ECMO
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Xiao Tang (Other)
Responsible Party: Sponsor-Investigator, Xiao Tang, Principal Investigator, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Other Study IDs: new anticoagulation of ECMO
Record Dates: First submitted 2018-04-04; First posted 2018-04-13 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Effective and normative anticoagulation is one of the most important components of Extracorporeal membrane oxygenation (ECMO) management. Excessive anticoagulation may lead to hemorrhage, which is the most common and serious complication. Currently, the most common factors for monitoring anticoagulation of ECMO are the activated clotting time (ACT) and activated partial thromboplastin time (APTT). However, there is a lack of a unified understanding of the related monitoring measures, monitoring targets, and bleeding risk assessments, which have been chosen mainly because of experiences reported by various ECMO centers or the results of retrospective studies.Therefore, anticoagulation strategies need to be improved. Our research have found ECMO anticoagulation management should be transformed from monitoring only the APTT/activated clotting time (ACT) to considering the entire coagulation process. To maintain thrombosis ability and PLT function within normal ranges may help reduce hemorrhage rates and improve prognoses. This randomized controlled study aim to develop the safety and efficacy new anticoagulation strategies of VV-ECMO.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years old, VV-ECMO is estimated more than 3 days

Exclusion Criteria:

* hemorrhage before VV-ECMO established, VV-ECMO more than 48 hours before admitted, VV-ECMO is estimated less than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients received ECMO support
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with hemorrhage events | 4 weeks
  1) fatal bleeding; 2) symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome; and/or 3. bleeding causing a drop in hemoglobin level by 20 g/L or more or requiring transfusion of two units of whole blood or red cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of respiratory and critical care medicine,Beijing Chao-yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided